CLINICAL TRIAL: NCT06197750
Title: Effect of Vestibular Stimulation on Motor Proficiency and Balance Among Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0745
Record Dates: First submitted 2023-02-05; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Vestibular System Disorder
Keywords: Vestibular stimulation (VeS); Hypotonic cerebral palsy
MeSH Terms: conditions — Vestibular Diseases; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular stimulation (Experimental): Group A received the vestibular stimulation by swing in different positions supine, prone and with or without support in each position for 10minnts 3 times a week for 10 weeks along with general strengthening exercises of upper and lower limb and
  Interventions: Other: Vestibular stimulation
- general strengthening exercises (Active Comparator): group B will receive general strengthening exercises of whole body for same time period.
  Interventions: Other: General strengthening exercises

INTERVENTIONS:
Other: Vestibular stimulation — Vestibular stimulation by swing
  Arms: Vestibular stimulation
Other: General strengthening exercises — General strengthening exercises
  Arms: general strengthening exercises

SUMMARY:
This was a randomized controlled trial study where there the total participants were 22and these participants were randomly selected and then distributed in to two groups all participants were selected according to the inclusion exclusion criteria of the study and then they were randomly distributed in two groups named as group A and group B both of the contain equal number of participants which are randomly distributed in groups each group contain 11 participants .Group A received the vestibular stimulation by swing in different positions supine, prone and with or without support in each position for 10minnts 3 times a week for 10 weeks along with general strengthening exercises of upper and lower limb and group B will receive general strengthening exercises of whole body for same time period. Data will be then analyzed by using SPSS windows version 25

DETAILED DESCRIPTION:
This was a randomized controlled trial study where there the total participants were 22and these participants were randomly selected and then distributed in to two groups all participants were selected according to the inclusion exclusion criteria of the study and then they were randomly distributed in two groups named as group A and group B both of the contain equal number of participants which are randomly distributed in groups each group contain 11 participants .Group A received the vestibular stimulation by swing in different positions supine, prone and with or without support in each position for 10minnts 3 times a week for 10 weeks along with general strengthening exercises of upper and lower limb and group B will receive general strengthening exercises of whole body for same time period.

ELIGIBILITY:
Inclusion Criteria:• Down syndrome

* Age 6 to 11 years
* Having no other medical history (6)

Exclusion Criteria:

* • Visual impairment

  * Patient with hearing impairment
  * Patient with poor cognition (6, 8)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 16 WEEKS
  Improvement in balance from baseline among children with Down syndrome
motor proficiency | 16 WEEKS
  Improvement in motor proficiency from baseline among children with Down syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Rabia Razzaq, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No